CLINICAL TRIAL: NCT06011642
Title: Reliability, Validity and Acceptance of the Kinder-eDIPS (Diagnostisches Interview Bei Psychischen Störungen im Kindes- Und Jugendalter)
Brief Title: Reliability and Validity of a Digital Version of a Structured Interview for Children and Adolescents (Kinder-eDIPS)
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Ruth von Brachel, Dr., Ruhr University of Bochum
Other Study IDs: 737
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Psychological Disease
Keywords: structured interview; psychological disease; children and adolescents

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clinical sample: Participants will be recruited from families in Bochum who receive treatment or wait for the treatment to begin at the Forschungs- und Behandlungszentrum (FBZ; outpatient treatment center).
  Interventions: Diagnostic Test: Diagnostisches Interview bei psychischen Störungen im Kindes- und Jugendalter, digitale Version (Kinder-eDIPS)
- Nonclinical sample: Participants will be recruited from families in Bochum who take part in experiments and studies at the Department of Clinical Child and Adolescent Psychology at the Ruhr-University. The Department of Clinical Child and Adolescent Psychology maintains a database of families interested in participating in research.
  Interventions: Diagnostic Test: Diagnostisches Interview bei psychischen Störungen im Kindes- und Jugendalter, digitale Version (Kinder-eDIPS)

INTERVENTIONS:
Diagnostic Test: Diagnostisches Interview bei psychischen Störungen im Kindes- und Jugendalter, digitale Version (Kinder-eDIPS) — The Kinder-eDIPS is a digital, structured interviews which assesses the most frequent psychological disorders. It exists in a parent and a child version. It can be delivered by trained clinicians and takes between 60 and 120 minutes.

SUMMARY:
The Kinder-eDIPS is a digital version of the Kinder-DIPS (Diagnostisches Interview bei Psychischen Störungen im Kindes- und Jugendalter), a structured interview to assess a variety of the most frequent psychological disorders in children and adolescents. In this study, the reliability, validity and acceptance of the Kinder-eDIPS will be tested in both a clinical and a non-clinical sample.

DETAILED DESCRIPTION:
The Kinder-eDIPS is a digital version of the Kinder-DIPS (Diagnostisches Interview bei Psychischen Störungen im Kindes- und Jugendalter), a structured interview to assess a variety of the most frequent psychological disorders in children and adolescents. The interview is administered by trained clinicians with children/adolescents and one of their primary carers. The reliability, validity and acceptance of former versions of the Kinder-DIPS (Kinder-DIPS for DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) and DSM-III) have been studied. The aim of the present study is to test the reliability, validity and acceptance of the newly developed digital version of the Kinder-DIPS, the Kinder-eDIPS, in both a clinical and a non-clinical sample.

ELIGIBILITY:
Inclusion Criteria:

* sufficient knowledge of the German language

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All families with children in the according age group who are willing to complete the structured interview and the questionnaires of the online-survey are allowed to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Kinder-eDIPS | within 1 week of the other measures
  digital, structured interview for children, adolescents and their parents/primary carers

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | within 1 week of the other measures
  Questionnaire assessing emotional symptoms,conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behaviour in 4-17 year olds (child and parent version)
Spence Children's Anxiety Scale (SCAS) | within 1 week of the other measures
  Questionnaire assessing anxiety symptoms in 7-17 year olds (child and parent version)
Short Mood and Feelings Questionnaire (SMFQ) | within 1 week of the other measures
  Questionnaire assessing depressive symptomology in 6-17 year olds (child and parent version)
Child and Adolescent Trauma Screening (CATS) | within 1 week of the other measures
  Questionnaire assessing potentially traumatic events and posttraumatic stress symptoms in 7-17 year olds (child and parent version)
Short form of the Eating Disorder Examination-Questionnaire adapted for children (ChEDE-Q8) | within 1 week of the other measures
  Questionnaire assessing eating disorder psychopathology in 7-18 year olds (only child version)

OTHER OUTCOMES:
Acceptance of the Interview | within 1 week of the other measures
  Questionnaire assessing children's/adolescent's and parent's perception of the interview

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Schneider, Prof., Study Director — Ruhr-University; Ruth von Brachel, Dr., Principal Investigator — Ruhr-University
Locations (1):
- Ruhr-University, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No